CLINICAL TRIAL: NCT03837028
Title: The Effect of Human Papilloma Virus Genotype on Women's Sexual Life
Brief Title: The Human Papilloma Virus Effect on Sexual Life
Acronym: HPVandFSFI
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: BakirkoyDr.SadiKonuk
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Results first posted 2020-09-01 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HPV 16/18 (+), cytology normal: Women who have HPV 16/18 positivity and normal cytology results in their cervical cancer screening test (co-test) results.
  The FSFI and BAI questionnaires were performed to the women in this group at the time of admission and two months later.
  Interventions: Other: FSFI
- HPV 16/18 (+), cytology abnormal: Women who have HPV 16/18 positivity and abnormal cytology results in their cervical cancer screening test (co-test) results. The FSFI and BAI questionnaires were performed to the women in this group at the time of admission and two months later.
  Interventions: Other: FSFI
- non-16/18 HPV (+), cytology abnormal: Women who have non- 16/18 high-risk HPV positivity and abnormal cytology results in their cervical cancer screening test (co-test) results. The FSFI and BAI questionnaires were performed to the women in this group at the time of admission and two months later.
  Interventions: Other: FSFI
- non-16/18 HPV (+), cytology normal: Women who have non- 16/18 high-risk HPV positivity and normal cytology results in their cervical cancer screening test (co-test) results. The FSFI and BAI questionnaires were performed to the women in this group at the time of admission and two months later.
  Interventions: Other: FSFI

INTERVENTIONS:
Other: FSFI — Sexual dysfunction was assessed via the self-administered Female Sexual Function Index Questionnaire which was adapted to the Turkish population. This is a 19-item questionnaire that covers six domains: desire; arousal, lubrication, orgasm, satisfaction, and pain. The full score is obtained by adding the six domain scores. FSFI scores range from 2.0 to 36.0, with higher scores indicating better sexual functioning.
  Other Names: Female Sexual Function Index Questionnaire

SUMMARY:
Human Papilloma Virus (HPV) is one of the most common causes of sexually transmitted diseases and its link with malignancies is well established, especially with anogenital tract cancers (cervical, vaginal, vulvar, anal cancers). HPV 16 and 18 are the most commonly isolated HPV types in cervical cancer, however not all infections with HPV 16 or 18 progress to cancer. After the HPV test has been used in cervical cancer screening, there have been concerns about whether women carry this virus. Although HPV testing may cause negative emotional responses, adverse emotional responses are related to HPV infection rather than testing. In this respect, there were several studies which evaluated the quality of life and psychological responses of women with positive HPV test results and it is known that positive HPV test results cause additional anxiety, distress and negative emotional responses in women. We hypothesized that the awareness of having a sexually transmitted infection in women with HPV and, therefore, a close follow-up and the need for further investigation such as colposcopy can affect their sexual life. In this study, we aimed to observe the changes in sexual function and anxiety of the HPV positive women with validated objective tools after being informed about their co-test results.

DETAILED DESCRIPTION:
The present prospective, observational study was undertaken among women who were attended to our gynecology outpatient clinic due to HPV positivity according to the cervical cancer screening programme. After the ethics approval was obtained from our hospital's local ethics committee, women aged between 30 and 50 years, sexually active, and who were first diagnosed with high risk HPV positive (HPV 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 68, 69, 82) were included in the study. Women with HPV positive were given standard information about HPV and HPV testing (co-test) developed by a clinical expert. This information includes; sexually transmitted nature of HPV, its high prevalence in sexually active women, usually transient nature of HPV, the association between high risk and low- risk HPV types and cervical intraepithelial neoplasia (CIN) and cervical cancer, the importance of HPV 16/18 positivity for cervical premalignant and malign lesions. After given the standard information, the patients were informed about their co-test results including HPV genotype, cytology results. The demographic data of the patients such as gravidity, parity,Body Mass Index (BMI), educational status, and marital status were recorded at the time of admission. The routine gynecologic examination was performed to all participants. The BMI was calculated as weight (kg) divided by the square of the height (m2). The patients were divided into four groups according to their HPV genotype and cytology results. The patients were divided into four groups according to their HPV genotype and cytology results. Group 1: HPV 16/18 (+), cytology normal, Group 2: HPV 16/18 (+), cytology abnormal, Group 3: non-16/18 HPV (+), cytology abnormal, Group 4: non-16/18 HPV (+), cytology normal. In our clinic, we manage the patients with abnormal co-test results according to the American Society for Colposcopy and Cervical Pathology guidelines. The patients in group 1, 2, and 3 were referred to colposcopy according to American Society for Colposcopy and Cervical Pathology (ASCCP) guideline and the patients in group 4 were referred to colposcopy according to their symptoms and vaginal examination results such as suspicious cervical observation for cervical intraepithelial neoplasia, postcoital bleeding and all of the participants were informed about the colposcopy procedure. All of the patients called for a follow-up visit two months later and were performed a colposcopy. Sexual function of the patients was assessed at the time of admission and two months later via the self-administered Female Sexual Function Index (FSFI) questionnaire. The anxiety status of the patients has assessed via the Beck Anxiety Inventory (BAI) questionnaire at the time of admission and 2 months later.

Cervical Cancer Screening and management of the results:

According to the national cervical cancer screening program in our country, screening is initiating at the age of 21 and women age <30 are screening with Papanicolaou test alone at intervals of every three years. Women ≥ 30 years have been screening with co-testing (HPV testing and Pap test) every five years. When HPV positivity is detected in the co-test, the HPV genotype is determined and the pap test is evaluated cytologically. While the patients with HPV 16/18 positive (cytology normal or abnormal) and non-HPV 16/18 positive and cytology abnormal referred to a specialist gynecologist for colposcopy, it is recommended that patients who have a non-HPV 16/18 positive and cytology normal should have a co-test after 1 year.

Beck Anxiety Inventory The Beck Anxiety Inventor (BAI) is a brief measure of anxiety with a focus on somatic symptoms of anxiety that was developed as a measure adept at discriminating between anxiety and depression. The BAI is administered via self-report and includes assessment of symptoms such as nervousness, dizziness, inability to relax, etc. The BAI has a total of 21 items. Respondents indicate how much they have been bothered by each symptom over the past week. Responses are rated on a 4-point Likert scale and range from 0 (not at all) to 3 (severely). The BAI is used in efforts to obtain a purer measure of anxiety that is relatively independent of depression. The total score is calculated by finding the sum of the 21 items. It is defined as; Score of 0-21 = low anxiety Score of 22-35 = moderate anxiety Score of 36 and above = potentially concerning levels of anxiety Female Sexual Function Index Sexual dysfunction was assessed via the self-administered FSFI which was adapted to the Turkish population. This is a 19-item questionnaire that covers six domains: desire (two questions); arousal and lubrication (four questions each); and orgasm, satisfaction, and pain (three questions each). The possible scores are 0-5 for the arousal, lubrication, orgasm, and pain domains; 1-5 for the satisfaction domain; and 1-5 for the desire domain. Domain scores were obtained by summing the scores of the individual items comprising the domain and then multiplying by the following domain factors: 0.6 for desire, 0.3 for arousal and lubrication, and 0.4 for orgasm, satisfaction, and pain. Regarding the individual domains, a score of less than 65% of the maximum achievable score was considered to indicate dysfunction in that domain. Thus, a score of less than 3.9 in each domain was considered to indicate Female sexual disorder (FSD). The full score is obtained by adding the six domain scores. FSFI scores range from 2.0 to 36.0, with higher scores indicating better sexual functioning. The total FSFI score was calculated and categorized as a dichotomous variable using 26.55 as a cutoff for overall Female sexual disorder. Sexual function was further categorized into four groups, as described previously: normal sexual function (total FSFI score ≥26.55), mild Female sexual disorder (total FSFI score 18-26.55), moderate Female sexual disorder (total FSFI score 11-17), and severe Female sexual disorder (total FSFI score ≤10).

We compared the FSFI and BAI scores between the groups and between the time of admission and 2 months later.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 30 and 50 years
* sexually active women
* women who were first diagnosed with high risk HPV positive (HPV 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 68, 69, 82)

Exclusion Criteria:

* postmenopausal women (defined as those with at least 12 consecutive months of amenorrhea with no other medical cause and a follicle- stimulating hormone (FSH) level of 40)
* women with chronic disease
* patients with antidepressant usage or patients with psychiatric disorders
* women who did not agree to participate in the study after reading the informed consent form
* women who admitted for follow up due to prior HPV infection
* women with only low-risk HPV (HPV 6, 11) positivity
* women with a sexual abuse history
* women with sexual penetration disorder

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who were attended to our gynecology outpatient clinic due to HPV positivity according to the cervical cancer screening programme were recruited in this study.
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Alay, Principal Investigator — University Of Health Sciences Bakirkoy Sadi Konuk Training And Research Hospital
Locations (1):
- Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The researchers in the study have not yet taken a decision on individual participant data (IPD) sharing.

RESULTS

PARTICIPANT FLOW:
Groups:
- Human Papillomavirus (HPV) 16/18 (+), Cytology Normal: Women who have Human papillomavirus (HPV) (16/18 positivity and normal cytology results in their cervical cancer screening test (co-test) results.
  The Female Sexual Function Index (FSFI) and Beck Anxiety Inventory (BAI) questionnaires were performed to the women in this group at the time of admission and two months later.
  FSFI: Sexual dysfunction was assessed via the self-administered FSFI Questionnaire which was adapted to the Turkish population. This is a 19-item questionnaire that covers six domains: desire; arousal, lubrication, orgasm, satisfaction, and pain. The full score is obtained by adding the six domain scores. FSFI scores range from 2.0 to 36.0, with higher scores indicating better sexual functioning.
- Human Papillomavirus (HPV)16/18 (+), Cytology Abnormal: Women who have HPV 16/18 positivity and abnormal cytology results in their cervical cancer screening test (co-test) results. The Female Sexual Function Index (FSFI) and Beck Anxiety Inventory (BAI) questionnaires were performed to the women in this group at the time of admission and two months later.
  FSFI: Sexual dysfunction was assessed via the self-administered FSFI Questionnaire which was adapted to the Turkish population. This is a 19-item questionnaire that covers six domains: desire; arousal, lubrication, orgasm, satisfaction, and pain. The full score is obtained by adding the six domain scores. FSFI scores range from 2.0 to 36.0, with higher scores indicating better sexual functioning.
- Non-16/18 Human Papillomavirus (HPV) (+), Cytology Abnormal: Women who have non- 16/18 high-risk HPV positivity and abnormal cytology results in their cervical cancer screening test (co-test) results. The Female Sexual Function Index (FSFI) and Beck Anxiety Inventory (BAI) questionnaires were performed to the women in this group at the time of admission and two months later.
  FSFI: Sexual dysfunction was assessed via the self-administered FSFI Questionnaire which was adapted to the Turkish population. This is a 19-item questionnaire that covers six domains: desire; arousal, lubrication, orgasm, satisfaction, and pain. The full score is obtained by adding the six domain scores. FSFI scores range from 2.0 to 36.0, with higher scores indicating better sexual functioning.
- Non-16/18 Human Papillomavirus (HPV) (+), Cytology Normal: Women who have non- 16/18 high-risk HPV positivity and normal cytology results in their cervical cancer screening test (co-test) results. The Female Sexual Function Index (FSFI) and Beck Anxiety Inventory (BAI) questionnaires were performed to the women in this group at the time of admission and two months later.
  FSFI: Sexual dysfunction was assessed via the self-administered FSFI Questionnaire which was adapted to the Turkish population. This is a 19-item questionnaire that covers six domains: desire; arousal, lubrication, orgasm, satisfaction, and pain. The full score is obtained by adding the six domain scores. FSFI scores range from 2.0 to 36.0, with higher scores indicating better sexual functioning.
Period: Overall Study
Arm/Group | Human Papillomavirus (HPV) 16/18 (+), Cytology Normal | Human Papillomavirus (HPV)16/18 (+), Cytology Abnormal | Non-16/18 Human Papillomavirus (HPV) (+), Cytology Abnormal | Non-16/18 Human Papillomavirus (HPV) (+), Cytology Normal
Started | 35 | 34 | 33 | 25
Completed | 19 | 23 | 20 | 18
Not Completed | 16 | 11 | 13 | 7
Not completed — Lost to Follow-up | 4 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 12 | 11 | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- HPV 16/18 (+), Cytology Normal: Women who have HPV 16/18 positivity and normal cytology results in their cervical cancer screening test (co-test) results.
  The FSFI and BAI questionnaires were performed to the women in this group at the time of admission and two months later.
  FSFI: Sexual dysfunction was assessed via the self-administered Female Sexual Function Index Questionnaire which was adapted to the Turkish population. This is a 19-item questionnaire that covers six domains: desire; arousal, lubrication, orgasm, satisfaction, and pain. The full score is obtained by adding the six domain scores. FSFI scores range from 2.0 to 36.0, with higher scores indicating better sexual functioning.
- Total: Total of all reporting groups
Arm/Group | HPV 16/18 (+), Cytology Normal | HPV 16/18 (+), Cytology Abnormal | Non-16/18 HPV (+), Cytology Abnormal | Non-16/18 HPV (+), Cytology Normal | Total
Number analyzed (Participants) | 19 | 23 | 20 | 18 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (5.6) | 37.7 (4.9) | 36.6 (4.8) | 40.1 (4.5) | 38.1 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 20 | 18 | 80
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Overall Female Sexual Function Index Score [Median (Full Range); unit: scores on a scale] — Female sexual function index (FSFI) covers six domains: desire, arousal, lubrication, and orgasm, satisfaction, and pain. The overall FSFI score is obtained by summing the six domain scores and ranges between 2.0 and 36.0, with higher scores indicating better sexual functioning. We presented the baseline overall FSFI score of the study groups in this section.
  scores on a scale | 25.2 [19.8 to 30.2] | 27.1 [16.6 to 35.6] | 23.8 [17.4 to 31.6] | 23 [15.3 to 34] | 25.1 [16.6 to 35.6]

OUTCOME MEASURES:

1. Primary Outcome: Female Sexual Function Index (FSFI) Score
Description: This is a 19-item questionnaire that covers six domains: desire, arousal, lubrication, and orgasm, satisfaction, and pain. The ranges of the domain scores are as follows: for desire 1.2 - 6.0, for arousal, lubrication, orgasm and pain 0 - 6.0 and for satisfaction 0.8 - 6.0. The higher scores of the six domains indicate better sexual functioning about that domain. The overall FSFI score is obtained by summing the six domain scores. The overall FSFI scores range from 2.0 to 36.0, with higher scores indicating better sexual functioning. The change between the initial and second months overall and six domain scores are our first primer outcomes.
Time Frame: change from initial overall FSFI score at second months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HPV 16/18 (+), Cytology Normal | HPV 16/18 (+), Cytology Abnormal | Non-16/18 HPV (+), Cytology Abnormal | Non-16/18 HPV (+), Cytology Normal
Number analyzed (Participants) | 19 | 23 | 20 | 18
score on a scale | 0.8 (0.5) | 1.2 (0.9) | 0.9 (0.9) | 0.7 (0.5)

2. Secondary Outcome: Beck Anxiety Inventory (BAI) Score
Description: The BAI has a total of 21 items. Respondents indicate how much they have been bothered by each symptom over the past week. Responses are rated on a 4-point Likert scale and range from 0 (not at all) to 3 (severely). The total score is calculated by finding the sum of the 21 items. The BAI scores range from 0 to 63 and higher scores are associated with high anxiety levels.
Time Frame: change from initial BAI score at second months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HPV 16/18 (+), Cytology Normal | HPV 16/18 (+), Cytology Abnormal | Non-16/18 HPV (+), Cytology Abnormal | Non-16/18 HPV (+), Cytology Normal
Number analyzed (Participants) | 19 | 23 | 20 | 18
score on a scale | 4.5 (3.0) | 4.8 (2.3) | 4.1 (2.1) | 2.2 (2.2)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | HPV 16/18 (+), Cytology Normal | HPV 16/18 (+), Cytology Abnormal | Non-16/18 HPV (+), Cytology Abnormal | Non-16/18 HPV (+), Cytology Normal
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/23 | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/23 | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/23 | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT03837028/Prot_SAP_000.pdf